CLINICAL TRIAL: NCT01672164
Title: Discovery and Validation of Proteogenomic Biomarker Panels in a Prospective Serial Blood and Urine Monitoring Study of Liver Transplant Recipients - Transplant Proteogenomics
Brief Title: Discovery and Validation of Proteogenomic Biomarker Panels in Liver Transplant Recipients
Acronym: PROGENI-LI
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOT-14
Record Dates: First submitted 2012-08-16; First posted 2012-08-24 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Liver Transplant Recipients; Liver Transplantation
Keywords: proteogenomic biomarker panels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma, serum, urine supernatant, urine pellet and tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Liver Transplant Recipients

SUMMARY:
The main focus of this study is to develop blood and/or urine tests that will help to detect early signs of rejection in people who have had a liver transplant. Researchers will examine blood, urine, and tissue samples and try to identify markers for certain conditions such as rejection, response to therapy, and scarring of the liver. Additionally, researchers would like to identify biomarkers that can detect damage to the native kidneys before blood levels of creatinine rises. By studying gene expression, researchers hope to be able to diagnose these conditions earlier and improve liver survival.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing primary deceased-donor or living donor liver transplantation;
* Subject must be able to understand and provide informed consent.

Exclusion Criteria:

* Need for combined organ transplantation;
* Previous solid organ and/or islet cell transplantation;
* Infection with HIV;
* Allergy to iodine;
* Inability or unwillingness of a participant to comply with study protocol;
* Any condition that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver Transplant Recipients
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Acute Rejection | 3 months after liver transplant
  The primary endpoint is the incidence of biopsy proven AR at 3, 12 and 24 months after LT.
Acute Rejection | 12 months after liver transplant
Acute Rejection | 24 months after liver transplant

SECONDARY OUTCOMES:
Severity of acute rejection | Baseline (Visit 1) to Month 24 (Visit 12):
  Severity (initial grade, steroid-responsive vs. refractory by biopsy) and clinical/biochemical resolution following treatment of AR
Recurrent Hepatitis-C Virus (HCV-R) | Baseline (Visit 1) to Month 24 (Visit 12)
  Incidence, severity (grade, stage), and treatment (requirement for, response rates) of HCV-R
Chronic Kidney Disease(CKD) | Baseline (Visit 1) to Month 24 (Visit 12)
  Incidence, severity (stage, need for renal replacement therapy or kidney transplantation), and response to treatment (CNI reduction/withdrawal ± MPA or mTOR) of CKD
Incidence of death, graft loss, and need for liver retransplantation | Baseline (Visit 1) to Month 24 (Visit 12)
Incidence of opportunistic infections, malignancy, and cardiovascular complications | Baseline (Visit 1) to Month 24 (Visit 12)
mRNA expression profiles of peripheral blood (AR, HCV-R, CKD) | Baseline (Visit 1) to Month 24 (Visit 12)
mRNA expression profiles of liver biopsies (AR, HCV-R) | Baseline (Visit 1) to Month 24 (Visit 12)
Protein expression profiles of plasma ( AR, HCV-R, CKD) | Baseline (Visit 1) to Month 24 (Visit 12)
Protein expression profiles of urine (CKD) | Baseline (Visit 1) to Month 24 (visit 12)
microRNA Profiling Plasma & Cells | Baseline (Visit 1) to Month 24 (Visit 12)
Multiparameter Flow Cytometry - Viral Pathogens | Baseline (Visit 1) to Month 24 (Visit 12)
Viral Monitoring - EBV & CMV | Baseline (Visit 1) to Month 24 (Visit 12)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Levitsky, MD, MS, Study Chair — Northwestern University Feinberg School of Medicine; Michael Abecassis, MD, MBA, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (6):
- United States (6):
  - Mayo Clinic, Phoenix, Arizona
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Mount Sinai School of Medicine, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data in ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools that are available to researchers who register online and subsequently receive DAIT approval.

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov
- See also: Clinical Trials in Organ Transplantation (CTOT) — http://www.ctotstudies.org/